CLINICAL TRIAL: NCT07028125
Title: Digital Monitoring of Self-reported Symptoms by Patients Treated With Cabozantinib Plus Nivolumab for Advanced Clear-cell Renal Carcinoma: The CANIQOL Multicentre Study
Brief Title: Digital Monitoring of Self-reported Symptoms by Patients Treated With Cabozantinib Plus Nivolumab for Advanced Clear-cell Renal Carcinoma
Acronym: CANIQOL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-518991-30-00; 2024-518991-30-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-10; First posted 2025-06-19 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Renal Cell Carcinoma (Kidney Cancer); Metastatic Renal Cell Carcinoma; Locally Advanced
Keywords: kidney cancer; metastatic; cabozantinib; nivolumab; digital monitoring system
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasm Metastasis | interventions — cabozantinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital monitoring under Cabozantinib and nivolumab treatments (Experimental): During this combined treatment, the digital monitoring system is used to collect weekly data on treatment tolerance by patient self-report.
  The digital telemonitoring platform is used to facilitate the monitoring of signs and symptoms of treatment-specific Adverse Events.
  The platform integrates an algorithm to define patient risk based on responses to data collected on platform.
  The self-reported information on the mobile digital device allows to "classify" patients ("correct", "compromised", "to be monitored", or "critical) and to create some alerts.
  Some actions may be undertaken depending on these alerts, with adjustments of the management of treatments
  Interventions: Drug: cabozantinib and nivolumab

INTERVENTIONS:
Drug: cabozantinib and nivolumab — cabozantinib and nivolumab according to the labelling indication, namely:
  * CABOZANTINIB 40 mg per oral route once daily
  * NIVOLUMAB 240 mg per intravenous route every 2 weeks
  During this combined treatment, the digital monitoring system is used to collect weekly data on treatment tolerance by patient self-report.

SUMMARY:
The aim of the study is to evaluate the impact of digital monitoring of self-reported symptoms (PROs) on the adjustment of treatment management in patients treated with cabozantinib plus nivolumab for advanced clear cell renal cell carcinoma (RCC) in real life during the first 3 months of combined treatment

DETAILED DESCRIPTION:
Patients receive the combination of Cabozantinib and Nivolumab as indicated in the label.

During this combined treatment, the digital monitoring system is used to collect weekly data on treatment tolerance, based on patient reports.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* Diagnosis of advanced/metastatic Renal Cell Carcinoma (RCC) with a clear-cell component
* No prior systemic treatment for RCC
* Physician-initiated decision prior to study enrollment to treat with cabozantinib and nivolumab in combination, in first line for advanced/metastatic RCC, according to approved local labels
* Female subjects of childbearing potential must not be pregnant at screening and during treatment by Cabozantinib and Nivolumab. Effective methods of contraception must be used throughout the course of treatment and for at least 5 months after the end of treatment. Sexually active fertile subjects and their partners must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the study and 5 months after the last dose of study treatment, even if oral contraceptives are also used.
* Subject affiliated to an appropriate social security system
* Patient has signed informed consents obtained before any trial related activities and according to local guidelines

Exclusion Criteria:

* Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol
* Current participation in another clinical study and/or in an investigational program with any intervention that could possibly interfere with the treatment and impact this study
* Patient with history of allergy or hypersensitivity to components of the study drugs
* Patient with contraindication to the study drugs
* Pregnant or lactating woman
* Patient unable to use digital tools
* Patient deprived of liberty or placed under the authority of a tutor
* Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with adjustment of treatments management | within the first 3 months of the combined treatment (cabozantinib and nivolumab)
  rate of patients with adjustment of treatments management including any unplanned action guided by weekly digital monitoring of self-reported symptoms: anticipated consultation, anticipated phone follow-up, anticipated advices, treatment discontinuation, hospitalization within the first 3 months of the combined treatment

SECONDARY OUTCOMES:
- The evolution of self-reported symptoms | during the first 6 months of the combination (cabozantinb and nivolumab)
  report regular follow-up of self-reported symptoms on the digital platform
- To evaluate the improvement of self-reported symptoms after adjustment of the combined treatment | during the first 3 months of the combination (cabozantinib and nivolumab)
  Follow-up of number of grade 3-4 of self-reported symptoms after modification of treatment management induced by remote follow-up at 3 months
- To characterize and evaluate regular follow-up of patients self-reported fatigue | During the first 6 months of combination (cabozantinib and nivolumab)
  Score of self-reported fatigue by the questionnaire Facit-F (score between 0 and 160)
- To have a longitudinal assessment of general health-related quality of life (QoL) | During the first 6 months of combination (cabozantinib and nivolumab)
  - The evolution of general health-related quality of life with the score of FSKI-10 questionnaire (score between 0 and 40)
- To assess the feasibility of regular follow-up of PROs in real life | At 3 and 6 months after initiation of combination (cabozantinib and nivolumab)
  The levels of satisfaction and difficulties encountered by patients using the digital monitoring with the French validated version of the self-questionnaire F-SUS System Usability Scale (score between 0 and 50)
- To characterize and describe warning adverse reactions | During the first 6 months of the combination (cabozantinib and nivolumab)
  - The characterization and description of warning adverse reactions that may require therapeutic adaptation
- To characterize alerts issued by digital monitoring | During the first 6 months of the combination (cabozantinib and nivolumab)
  Follow-up of number of alerts issued by digital monitoring
To have a longitudinal assessment of anxiety/depression and pain | During the first 6 months of combination (cabozantinib and nivolumab)
  The evolution of anxiety/depression with HADS scale (score between 0 and 56)
To characterize alerts issued by digital monitoring | During the first 6 months of combination (cabozantinib and nivolumab)
  Follow-up on the type of alerts (dose adjustment or treatment discontinuation)

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Centre Hospitalier d'Annecy, Annecy
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de Bayeux, Bayeux
  - Centre François Baclesse, Caen
  - Polyclinique du Parc Elsan, Caen
  - Ghpso Creil, Creil
  - Centre Hospitalier de Lorient, Lorient
  - GHR Mulhouse Sud Alsace, Mulhouse
  - CHU, Saint-Etienne
  - Centre Hospitalier de Tours, Tours

IPD SHARING:
Plan to Share IPD: No